CLINICAL TRIAL: NCT00001597
Title: Pain Measurement in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970104; 97-D-0104
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Healthy; Pain
Keywords: Psychophysics; Validation; Fentanyl; Normal Volunteer; Pain
MeSH Terms: conditions — Pain

SUMMARY:
This study will attempt to develop and validate improved subjective measures of pain sensation and use these measures to evaluate pain sensitivity in patients.

Normal healthy volunteers and dental patients undergoing third molar extraction may be eligible for this study. Participants will undergo the following procedures:

Volunteers: Volunteers will participate in two 90-minute sessions in which they will receive and rate four heat stimuli per minute applied to the skin for a maximum of 36 minutes. The heat stimuli range from 37° (Degree)C to 51° (Degree)C (99° (Degree) F to 124° (Degree) F) and last 2 to 3 seconds. A drug commonly used in dental treatments may be administered during the second session. This will be either a maximum of 0.15 mg fentanyl, a short-acting narcotic pain killer, or a maximum of 5 mg saline, an inactive substance (placebo).

Dental patients: Dental patients will participate in two 60-minute sessions. The first session will be on the day before the third molar extraction, and the second session will be immediately before the dental procedure. The heat stimulus procedure will be identical to that described above for normal healthy volunteers.

DETAILED DESCRIPTION:
Mismanaged pain is still a major medical problem. Many pain syndromes have no effective treatment, and many are managed poorly. Basic and applied research on pain treatment is hampered by the unobservable nature of pain sensation and the lack of validated measures of this perception.

The purpose of this protocol is to develop and validate improved subjective measures of pain sensation and use these measures to evaluate pain sensitivity in clinical populations. Normal volunteers rate experimentally-evoked pain sensations before and after double-blind administration of the opioid fentanyl or saline placebo. Patients rate experimentally-evoked pain sensations without any drug administration.

ELIGIBILITY:
Normal Volunteers, including NIH employees, will serve as subjects.

No subjects with any painful disease or diseases in which altered pain sensitivity is suspected.

No subjects will be included with poor general health, history of significant illness, history of psychotic disorder or recent emotional distress, serious heart, lung, or liver disease, or pregnancy.

Subjects also will be excluded on the basis of history of allergy to any of the medications, history of chronic or recent drug use that may alter pain response, or chronic drug abuse.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1997-03; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Gracely RH, McGrath P, Dubner R. Validity and sensitivity of ratio scales of sensory and affective verbal pain descriptors: manipulation of affect by diazepam. Pain. 1978 Jun;5(1):19-29. doi: 10.1016/0304-3959(78)90021-0. PMID 673439
- [Background] Gracely RH, Dubner R, McGrath PA. Narcotic analgesia: fentanyl reduces the intensity but not the unpleasantness of painful tooth pulp sensations. Science. 1979 Mar 23;203(4386):1261-3. doi: 10.1126/science.424753.
- [Background] Cannon RO 3rd, Quyyumi AA, Mincemoyer R, Stine AM, Gracely RH, Smith WB, Geraci MF, Black BC, Uhde TW, Waclawiw MA, et al. Imipramine in patients with chest pain despite normal coronary angiograms. N Engl J Med. 1994 May 19;330(20):1411-7. doi: 10.1056/NEJM199405193302003. PMID 8159194